CLINICAL TRIAL: NCT06260306
Title: Comparison of a Hip Activation Versus a Combined Hip Activation and Core Stabilization Program on Improving Lower Extremity Function: A Single-Blind Randomized Controlled Trial
Brief Title: Hip Activation vs. Hip Activation + Core Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002568
Record Dates: First submitted 2024-01-19; First posted 2024-02-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Movement, Abnormal; Lower Extremity Problem
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The PI who will be performing the data analysis will be blinded to participants' random group allocation. The other investigators who will be collecting the outcome data will know the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Activation Group (Active Comparator): The hip activation HEP group will receive a combination of hip musculature activation exercises used by previous researchers that show an increase in hip muscle recruitment.
  Interventions: Other: Hip activation home exercise program
- Combined Hip Activation and Core Stabilization Group (Experimental): The hip activation plus core stabilization HEP group will receive the same hip exercises as the other group, plus core stabilization exercises used by previous researchers.
  Interventions: Other: Hip activation plus core stabilization home exercise program

INTERVENTIONS:
Other: Hip activation home exercise program — The hip activation HEP group will receive a combination of hip musculature activation exercises used by previous researchers that show an increase in hip muscle recruitment. Each participant will perform their respective intervention program at home twice weekly for eight weeks.
  Arms: Hip Activation Group
Other: Hip activation plus core stabilization home exercise program — The hip activation plus core stabilization HEP group will receive the same hip exercises, plus core stabilization exercises used by previous researchers. Each participant will perform their respective intervention program at home twice weekly for eight weeks.
  Arms: Combined Hip Activation and Core Stabilization Group

SUMMARY:
The purpose of this investigation is to compare the effects of a combined hip activation and core stabilization training home exercise program (HEP) versus a hip activation training HEP alone on lower extremity (LE) frontal plane mechanics in healthy individuals.

Specific Aim 1: To determine whether between- and/or within-group differences exist on the Forward Step-Down test (FSDT) when comparing a combined hip activation and core stabilization training HEP as compared to a hip activation training HEP.

Specific Aim 2: To determine whether between- and/or within-group differences exist on the peak external knee abduction moment when comparing a combined hip activation and core stabilization training HEP to a hip activation training HEP.

Specific Aim 3: To determine whether between- and/or within-group differences exist on gluteal and core muscle surface electromyography (sEMG) when comparing a combined hip activation and core stabilization training HEP to a hip activation training HEP.

Specific Aim 4: To determine whether a dose-response relationship exists between HEP compliance and change on the FSDT, peak external knee abduction moment, and sEMG.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be current first- or second-year Doctor of Physical Therapy (DPT) students in the School of Allied Health Professions (SAHP) at Louisiana State University Health Shreveport over the age of 21.

Exclusion Criteria:

* Current pain or pathology in either LE which currently limits their ability to perform the FSDT or drop landing task, a history of low back pain in the last three months, known pregnancy, as pregnancy is a risk factor for diastasis rectus abdominis (DRA) which may be exacerbated by participation in the intervention and could be a confounding variable, and current participation in other clinical trials.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Forward Step Down Test (FSDT) | Pre- and post-eight week intervention
  Rating on the FSDT (0-6; 0-1 = good movement quality, 2-3 = moderate movement quality, 4 or more = poor movement quality).

SECONDARY OUTCOMES:
Maximal volitional isometric contraction (MVIC) via sensory electromyography (sEMG) of gluteus maximus (GMax) | Pre- and post-eight week intervention
  MVIC (microvolts) of GMax during performance of the FSDT
Mean activation of GMax via sEMG | Pre- and post-eight week intervention
  Mean activation (% MVIC) of GMax during performance of the FSDT
Peak activation of GMax via sEMG | Pre- and post-eight week intervention
  Peak activation (%MVIC) of GMax during performance of the FSDT
MVIC via sEMG of gluteus medius (GMed) | Pre- and post-eight week intervention
  MVIC (microvolts) of GMed during performance of the FSDT
Mean activation of GMed via sEMG | Pre- and post-eight week intervention
  Mean activation (% MVIC) of GMed during performance of the FSDT
Peak activation of GMed via sEMG | Pre- and post-eight week intervention
  Peak activation (% MVIC) of GMed during performance of the FSDT
MVIC via of transversus abdominis (TA) | Pre- and post-eight week intervention
  MVIC (microvolts) of TA during performance of the FSDT
Mean activation of TA via sEMG | Pre- and post-eight week intervention
  Mean activation (% MVIC) of TA during performance of the FSDT
Peak activation of TA via sEMG | Pre- and post-eight week intervention
  Peak activation (% MVIC) of TA during performance of FSDT
Peak external knee abduction moment during drop landing task | Pre- and post-eight week intervention
  Kinetic assessment of the peak external knee abduction moment (Nm/kg) during the drop landing task
Compliance with Home Exercise Program | Post-eight week intervention
  Self-reported completion of each HEP session will be recorded by the participant and then returned to the investigators post-completion

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Flowers, PT, DPT, PhD, Principal Investigator — LSU Health Sciences Center at Shreveport
Locations (1):
- LSU Health Sciences Center at Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark L, Dean A, Mitchell A, & Torgerson DJ. Envelope use and reporting in randomised controlled trials: a guide for researchers. Research Methods in Medicine & Health Sciences. 2021;2(1):2-11. doi:10.1177/2632084320957204
- [Background] Konrad P. The ABC of EMG: A Practical Introduction to Kinesiological Electromyography. Noraxon U.S.A.; 2006.
- [Result] Gage BE, McIlvain NM, Collins CL, Fields SK, Comstock RD. Epidemiology of 6.6 million knee injuries presenting to United States emergency departments from 1999 through 2008. Acad Emerg Med. 2012 Apr;19(4):378-85. doi: 10.1111/j.1553-2712.2012.01315.x. PMID 22506941
- [Result] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Result] Bolgla LA, Boling MC, Mace KL, DiStefano MJ, Fithian DC, Powers CM. National Athletic Trainers' Association Position Statement: Management of Individuals With Patellofemoral Pain. J Athl Train. 2018 Sep;53(9):820-836. doi: 10.4085/1062-6050-231-15. PMID 30372640
- [Result] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Result] Mascal CL, Landel R, Powers C. Management of patellofemoral pain targeting hip, pelvis, and trunk muscle function: 2 case reports. J Orthop Sports Phys Ther. 2003 Nov;33(11):647-60. doi: 10.2519/jospt.2003.33.11.647. PMID 14669960
- [Result] Leetun DT, Ireland ML, Willson JD, Ballantyne BT, Davis IM. Core stability measures as risk factors for lower extremity injury in athletes. Med Sci Sports Exerc. 2004 Jun;36(6):926-34. doi: 10.1249/01.mss.0000128145.75199.c3. PMID 15179160
- [Result] Huxel Bliven KC, Anderson BE. Core stability training for injury prevention. Sports Health. 2013 Nov;5(6):514-22. doi: 10.1177/1941738113481200. PMID 24427426
- [Result] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Result] Flowers DW, Brewer W, Mitchell K, Ellison J, Frilot C. The Effect of Core Stabilization Training on Improving Gait and Self-Perceived Function in Patients with Knee Osteoarthritis: A Single-Arm Clinical Trial. Pathophysiology. 2022 Sep 1;29(3):495-506. doi: 10.3390/pathophysiology29030040. PMID 36136067
- [Result] McCallister E, Flowers D. Can the Forward-Step-Down Test Be Used Reliably in the Clinical Setting to Assess Movement Changes Resulting from Maximal Exertion? A Pilot Study. Internet Journal of Allied Health Sciences and Practice. Published online 2020. doi:https://doi.org/10.46743/1540-580x/2020.1931
- [Result] Flowers DW, Brewer W, Ellison J, Mitchell K, Frilot C. Transversus abdominis activation does not alter gait impairments in patients with and without knee osteoarthritis. Clin Biomech (Bristol). 2021 Feb;82:105270. doi: 10.1016/j.clinbiomech.2020.105270. Epub 2021 Jan 1. PMID 33421757
- [Result] Cannon J, Weithman BA, Powers CM. Activation training facilitates gluteus maximus recruitment during weight-bearing strengthening exercises. J Electromyogr Kinesiol. 2022 Apr;63:102643. doi: 10.1016/j.jelekin.2022.102643. Epub 2022 Feb 9. PMID 35189569
- [Result] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582
- [Result] Park KM, Cynn HS, Choung SD. Musculoskeletal predictors of movement quality for the forward step-down test in asymptomatic women. J Orthop Sports Phys Ther. 2013;43(7):504-10. doi: 10.2519/jospt.2013.4073. Epub 2013 Jun 11. PMID 23756380
- [Result] Ishida T, Koshino Y, Yamanaka M, Ueno R, Taniguchi S, Samukawa M, Saito H, Matsumoto H, Aoki Y, Tohyama H. The effects of a subsequent jump on the knee abduction angle during the early landing phase. BMC Musculoskelet Disord. 2018 Oct 20;19(1):379. doi: 10.1186/s12891-018-2291-4. PMID 30342498
- [Result] McNair PJ, Prapavessis H. Normative data of vertical ground reaction forces during landing from a jump. J Sci Med Sport. 1999 Mar;2(1):86-8. doi: 10.1016/s1440-2440(99)80187-x. PMID 10331479
- [Result] Argent R, Daly A, Caulfield B. Patient Involvement With Home-Based Exercise Programs: Can Connected Health Interventions Influence Adherence? JMIR Mhealth Uhealth. 2018 Mar 1;6(3):e47. doi: 10.2196/mhealth.8518. PMID 29496655
- [Result] Cavalli M, Aiolfi A, Bruni PG, Manfredini L, Lombardo F, Bonfanti MT, Bona D, Campanelli G. Prevalence and risk factors for diastasis recti abdominis: a review and proposal of a new anatomical variation. Hernia. 2021 Aug;25(4):883-890. doi: 10.1007/s10029-021-02468-8. Epub 2021 Aug 6. PMID 34363190
- [Result] Selkowitz DM, Beneck GJ, Powers CM. Which exercises target the gluteal muscles while minimizing activation of the tensor fascia lata? Electromyographic assessment using fine-wire electrodes. J Orthop Sports Phys Ther. 2013 Feb;43(2):54-64. doi: 10.2519/jospt.2013.4116. Epub 2012 Nov 16. PMID 23160432
- [Result] Harput G, Ulusoy B, Akmese R, Ergun N. Comparison of muscle activation levels and knee valgus between individuals with medial patellofemoral ligament reconstruction and healthy individuals during fatiguing step down task. Clin Biomech (Bristol). 2020 Aug;78:105067. doi: 10.1016/j.clinbiomech.2020.105067. Epub 2020 Jun 6. PMID 32535475
- [Result] Selkowitz DM, Beneck GJ, Powers CM. Comparison of Electromyographic Activity of the Superior and Inferior Portions of the Gluteus Maximus Muscle During Common Therapeutic Exercises. J Orthop Sports Phys Ther. 2016 Sep;46(9):794-9. doi: 10.2519/jospt.2016.6493. Epub 2016 Aug 5. PMID 27494053
- [Result] Okubo Y, Kaneoka K, Imai A, Shiina I, Tatsumura M, Izumi S, Miyakawa S. Electromyographic analysis of transversus abdominis and lumbar multifidus using wire electrodes during lumbar stabilization exercises. J Orthop Sports Phys Ther. 2010 Nov;40(11):743-50. doi: 10.2519/jospt.2010.3192. PMID 21041966
- [Result] Fan B, Xia H, Xu J, Li Q, Shull PB. IMU-based knee flexion, abduction and internal rotation estimation during drop landing and cutting tasks. J Biomech. 2021 Jul 19;124:110549. doi: 10.1016/j.jbiomech.2021.110549. Epub 2021 Jun 13. PMID 34167019

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT06260306/Prot_SAP_000.pdf